CLINICAL TRIAL: NCT02384083
Title: Phase I/II, Multicenter, Open Label, Clinical Trial of Filanesib (ARRY-520) in Combination With Pomalidomide and Dexamethasone for Relapsed/Refractory (R/R) Multiple Myeloma (MM) Patients
Brief Title: Filanesib (ARRY-520) in Combination With Pomalidomide and Dexamethasone for Relapsed/Refractory (R/R) Multiple Myeloma (MM) Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Collaborators: Array BioPharma (Industry); Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: POMDEFIL
Record Dates: First submitted 2015-03-01; First posted 2015-03-10 (Estimated); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Pethema; Filanesib; Pomalidomide
MeSH Terms: conditions — Multiple Myeloma | interventions — filanesib; pomalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Filanesib, pomalidomide and dexamethasone (Experimental): 28-day cycles of Filanesib administered iv as a 1-hour (± 10-minute) infusion at escalating doses on days 1, 2, 15 & 16, + pomalidomide administered p.o. at escalating doses during 21 days with 7 days rest period + dexamethasone at a fixed dose of 40 mg po days 1, 8, 15 & 22
  Interventions: Drug: Filanesib, pomalidomide and dexamethasone

INTERVENTIONS:
Drug: Filanesib, pomalidomide and dexamethasone — Patients will be treated with 28-day cycles of Filanesib administered iv as a 1-hour (± 10-minute) infusion at escalating doses on days 1, 2, 15 & 16, + pomalidomide administered p.o. at escalating doses during 21 days with 7 days rest period + dexamethasone at a fixed dose of 40 mg po days 1, 8, 15 & 22. G-CSF prophylaxis is mandatory in all patients after Filanesib, starting from Day 3 and Day 17 (for a total of 7 days each). Treatment will be continued until progression or unacceptable toxicity.

SUMMARY:
Phase I/II, Multicenter, Open Label, Clinical Trial to evaluate safety and efficacy and determine the Maximum Tolerated Dose (MTD) of Filanesib in combination with pomalidomide and dexamethasone in relapsed/refractory (R/R) Multiple Myeloma (MM) patients

DETAILED DESCRIPTION:
National, multicenter, open label single-arm, non-comparative study, that will evaluate the MTD and the efficacy of the Kinesin Spindle Protein (KSP) inhibitor Filanesib (ARRY-520) in combination with pomalidomide + dexamethasone in relapsed or refractory MM patients.

For this purpose, relapsed or refractory MM patients after at least two prior lines of therapy including bortezomib and lenalidomide, who are refractory or intolerant to lenalidomide and refractory to the last line of therapy will be treated with 28-day cycles of Filanesib administered iv as a 1-hour (± 10-minute) infusion at escalating doses on days 1, 2, 15 & 16, + pomalidomide administered po at escalating doses during 21 days with 7 days rest period + dexamethasone at a fixed dose of 40 mg po days 1, 8, 15 & 22. G-CSF prophylaxis is mandatory in all patients after Filanesib, starting from Day 3 and Day 17 (for a total of 7 days each). Treatment will be continued until progression or unacceptable toxicity.

Initially, a Phase I will be conducted using a modified 3+3 dose-escalating algorithm. The first three patients will be enrolled in the first dose level (see Figure 1 for dose escalation levels). If no DLT occurs among them, the next cohort of three patients will continue at the next higher dose level. If a DLT occurs among the first three evaluable patients during the first cycle, three more patients will be enrolled at the same dose level.

If no more than one DLT is observed among the six evaluable patients in this expanded dose group during cycle 1, enrollment will continue at the next higher dose level following the same scheme.

If more than one DLT occurs among the three or six evaluable patients included in the 1st cohort, an alternative dose escalation will be started, with a reduction of the dose of pomalidomide (see Figure 1). Patients will be then treated following again the same 3+3 algorithm. If more than one DLT out of three or six patients occur at the first dose level of the alternative escalation, the study will be stopped.

MTD will be considered as the dose level in which ≤1 DLT are observed among 6 evaluable patients, therefore, at least six patients must be treated at a given dose before this dose is considered the MTD.

Once the MTD is determined in Phase I, additional patients will be treated at this dose in the Phase II portion of the trial in order to define the activity and further define the toxicity of the combination at the MTD.

Patient participation in the study will comprise several periods:

The pre-treatment period includes the screening visit. After providing the written Informed Consent form to participate in the study, patients will be evaluated for eligibility during a screening period of up to 21 days (Days -21 to -1).

During the treatment period, all patients will receive Filanesib in combination with pomalidomide and dexamethasone in 28-days-cycles until progression or unacceptable toxicity.

Patients receiving the combination will be evaluated for efficacy and toxicity after the completion of each cycle.

No intra-patient escalation will be performed, that is, patients included at a given dose level during the Phase I will remain at this dose level during all treatment unless a dose reduction is required for toxicity.

All patients that discontinue treatment for any other cause different to disease progression will be evaluated in the follow-up period every two months for 1 additional year, for disease status, survival and safety (including second primary malignancies). All patients that have progressed at the end of treatment will be followed for survival and safety only (including second primary malignancy), being phone contact acceptable.

Patients will be considered to be on-study from the signature of the Informed Consent to the end of the follow-up period. Patients will be considered to be on-treatment for the duration of their treatment and in the first 30 days following treatment discontinuation. Treatment discontinuation is defined as the day of the last study drug dose administration.

Patients will receive the study combination while it is considered to be in their best interest. Specifically, treatment will continue until one or more of the following events occur:

* Disease progression.
* Unacceptable toxicity.
* Patient refusal.
* Intercurrent serious illness.
* Protocol deviation with an effect on the risk/benefit ratio of the clinical trial.
* Treatment delay > 4 weeks (except in case of clear clinical benefit, with the sponsors' approval).
* Study closure.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Performance status (ECOG) ≤ 2.
* Patient is, in the Investigator's opinion, willing and able to comply with the protocol requirements.
* Patient has given voluntary written Informed Consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care.
* Patients previously diagnosed with MM according to the IMWG Criteria (Blood 2011) that after previous treatment with at least 2 regimens require therapy due to a relapse/progression of the disease.
* Regarding the disease history, patient must:

  * Have received 2 prior lines of therapy including bortezomib and lenalidomide.
  * Be refractory or intolerant to lenalidomide.
  * Be refractory to the last line of therapy.
  * Refractoriness to any therapy is defined as either failure to achieve minimal response with it, or development of progressive disease (PD) while on therapy or within 60 days after finishing it.
  * At least two cycles of treatment must have been received, unless PD is documented earlier.
* Only for the Phase II, patients must have measurable disease, defined as any of the following:

  * Serum monoclonal protein value ≥ 500 mg/dl.
  * Urine light chain excretion ≥ 200 mg/24 hours.
  * Abnormal serum free light chains (FLCs) ratio plus involved FLC level ≥ 10 mg/dl.

Exclusion Criteria:

* Prior therapy with Filanesib or pomalidomide.
* Non-adequate hematological or biochemical parameters as specified below:
* Hemoglobin < 8.0 g/dl.
* Platelets count < 75 x109/L without previous platelet transfusions in the last 7 days. If high bone marrow infiltration (>50%) is present, ≥ 50 x109/L platelet count is required.
* Neutrophils (ANC) <1.5 × 109/L without growth factor support (defined as no growth factor administration for at least 14 days prior to observation). If the bone marrow contains ≥ 50% plasma cells, a neutrophil count ≥1.0 × 109/L is allowed.
* Aspartate transaminase (AST): > 2.5 x the upper limit range.
* Alanine transaminase (ALT): > 2.5 x the upper limit range.
* Total bilirubin: > 2 x the upper limit range.
* Creatinine clearance: < 45 mL/min (measured or calculated with the Cockcroft and Gault formula).
* Absence of recovery from any significant non-hematological toxicity derived from previous treatments. The presence of alopecia and NCI-CTC grade < 2 symptomatic peripheral neuropathy is allowed.
* Concomitant anti-myeloma therapy, including corticosteroids at a dose greater than 10 mg/d prednisone or equivalent, within 14 days prior to Day 1 of Cycle 1.
* Pregnant or lactating women; men and women of reproductive potential who are not using highly effective contraceptive methods.
* Previous history of any other malignancy in the last five years (except basal cell carcinoma, skin epithelioma or carcinoma in situ of any site).
* Prior allogeneic bone marrow transplantation in the six prior months or active GVHD in the past month prior to cycle 1, day 1.
* Other relevant diseases or adverse clinical conditions:
* Congestive heart failure or unstable angina pectoris, myocardial infarction within 12 months before inclusion in the study.
* Uncontrolled arterial hypertension or unstable cardiac arrhythmias (i.e. requiring a change in medication within the last 3 months or a hospital admission within the past 6 months).
* History of significant neurological or psychiatric disorders.
* Active infection.
* Significant non-neoplastic liver disease (e.g., cirrhosis, active chronic hepatitis).
* Uncontrolled endocrine diseases (e.g. diabetes mellitus, hypothyroidism or hyperthyroidism) (i.e. requiring relevant changes in medication within the last month, or hospital admission within the last 3 months).
* Patient is known to be human immunodeficiency virus (HIV) positive, Hepatitis B surface antigen-positive or active hepatitis C infection.
* Limitation of the patient's ability to comply with the treatment or follow-up protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2020-03-23 (Actual)

PRIMARY OUTCOMES:
Maxim Tolerability Dose measured by common toxicity criteria v4.0 | 6 months

SECONDARY OUTCOMES:
Eficcacy measured by the rate of responses | 6 months
  Efficacy of the Kinesin Spindle Protein (KSP) inhibitor Filanesib (ARRY-520) in combination with pomalidomide + dexamethasone in relapsed or refractory MM patients.

CONTACTS AND LOCATIONS:
Overall Officials: Ocio Enrique, DR, Principal Investigator — PETHEMA Foundation
Locations (10):
- Spain (10):
  - Instoitut Català d'Oncologia, Badalona
  - Hospital Clinico Universitario, Barcelona
  - Hospital Doce de Octubre, Madrid
  - Hospital Morales Messeguer, Murcia
  - Clínica Universitaria de Navarra, Pamplona
  - Hospital Clinico Universitario Salamanca, Salamanca
  - Hospital General de Segovia, Segovia
  - Hospital Virgen del Rocío, Seville
  - Hospital Universitario Dr Peset, Valencia
  - Hospital Lozano Blesa, Zaragoza

REFERENCES:
- [Background] Kyle RA, Rajkumar SV. Multiple myeloma. N Engl J Med. 2004 Oct 28;351(18):1860-73. doi: 10.1056/NEJMra041875. No abstract available. PMID 15509819
- [Background] Kyle RA, Rajkumar SV. Multiple myeloma. Blood. 2008 Mar 15;111(6):2962-72. doi: 10.1182/blood-2007-10-078022. PMID 18332230
- [Background] Kumar SK, Lee JH, Lahuerta JJ, Morgan G, Richardson PG, Crowley J, Haessler J, Feather J, Hoering A, Moreau P, LeLeu X, Hulin C, Klein SK, Sonneveld P, Siegel D, Blade J, Goldschmidt H, Jagannath S, Miguel JS, Orlowski R, Palumbo A, Sezer O, Rajkumar SV, Durie BG; International Myeloma Working Group. Risk of progression and survival in multiple myeloma relapsing after therapy with IMiDs and bortezomib: a multicenter international myeloma working group study. Leukemia. 2012 Jan;26(1):149-57. doi: 10.1038/leu.2011.196. Epub 2011 Jul 29. PMID 21799510
- [Background] Ocio EM, Richardson PG, Rajkumar SV, Palumbo A, Mateos MV, Orlowski R, Kumar S, Usmani S, Roodman D, Niesvizky R, Einsele H, Anderson KC, Dimopoulos MA, Avet-Loiseau H, Mellqvist UH, Turesson I, Merlini G, Schots R, McCarthy P, Bergsagel L, Chim CS, Lahuerta JJ, Shah J, Reiman A, Mikhael J, Zweegman S, Lonial S, Comenzo R, Chng WJ, Moreau P, Sonneveld P, Ludwig H, Durie BG, Miguel JF. New drugs and novel mechanisms of action in multiple myeloma in 2013: a report from the International Myeloma Working Group (IMWG). Leukemia. 2014 Mar;28(3):525-42. doi: 10.1038/leu.2013.350. Epub 2013 Nov 20. PMID 24253022
- [Background] Mateos MV, Ocio EM, San Miguel JF. Novel generation of agents with proven clinical activity in multiple myeloma. Semin Oncol. 2013 Oct;40(5):618-33. doi: 10.1053/j.seminoncol.2013.07.005. PMID 24135407
- [Background] Miguel JS, Weisel K, Moreau P, Lacy M, Song K, Delforge M, Karlin L, Goldschmidt H, Banos A, Oriol A, Alegre A, Chen C, Cavo M, Garderet L, Ivanova V, Martinez-Lopez J, Belch A, Palumbo A, Schey S, Sonneveld P, Yu X, Sternas L, Jacques C, Zaki M, Dimopoulos M. Pomalidomide plus low-dose dexamethasone versus high-dose dexamethasone alone for patients with relapsed and refractory multiple myeloma (MM-003): a randomised, open-label, phase 3 trial. Lancet Oncol. 2013 Oct;14(11):1055-1066. doi: 10.1016/S1470-2045(13)70380-2. Epub 2013 Sep 3. PMID 24007748
- [Background] Ocio EM, Mitsiades CS, Orlowski RZ, Anderson KC. Future agents and treatment directions in multiple myeloma. Expert Rev Hematol. 2014 Feb;7(1):127-41. doi: 10.1586/17474086.2014.858595. Epub 2013 Dec 18. PMID 24350987
- [Background] Blangy A, Lane HA, d'Herin P, Harper M, Kress M, Nigg EA. Phosphorylation by p34cdc2 regulates spindle association of human Eg5, a kinesin-related motor essential for bipolar spindle formation in vivo. Cell. 1995 Dec 29;83(7):1159-69. doi: 10.1016/0092-8674(95)90142-6. PMID 8548803
- [Background] Stern BM, Murray AW. Lack of tension at kinetochores activates the spindle checkpoint in budding yeast. Curr Biol. 2001 Sep 18;11(18):1462-7. doi: 10.1016/s0960-9822(01)00451-1. PMID 11566107
- [Background] Tunquist BJ, Woessner RD, Walker DH. Mcl-1 stability determines mitotic cell fate of human multiple myeloma tumor cells treated with the kinesin spindle protein inhibitor ARRY-520. Mol Cancer Ther. 2010 Jul;9(7):2046-56. doi: 10.1158/1535-7163.MCT-10-0033. Epub 2010 Jun 22. PMID 20571074
- [Background] Boiani M, Daniel C, Liu X, Hogarty MD, Marnett LJ. The stress protein BAG3 stabilizes Mcl-1 protein and promotes survival of cancer cells and resistance to antagonist ABT-737. J Biol Chem. 2013 Mar 8;288(10):6980-90. doi: 10.1074/jbc.M112.414177. Epub 2013 Jan 22. PMID 23341456
- [Background] Lonial S, Shah JJ, Zonder J, Bensinger WI, Cohen AD, Kaufman JL, et al. Prolonged Survival and Improved Response Rates With ARRY-520 In Relapsed/Refractory Multiple Myeloma (RRMM) Patients With Low α-1 Acid Glycoprotein (AAG) Levels: Results From a Phase 2 Study. Blood. 2013;122(21):285-
- [Background] Shah JJ, Thomas S, Weber DM, Wang M, Orlowski R. Phase 1 Study Of The Novel Kinesin Spindle Protein Inhibitor Arry-520 + Carfilzomib(Car) In Patients With Relapsed And/Or Refractory Multiple Myeloma (RRMM). Haematologica. 2013;98(S1):Abstract-S579
- [Background] Humphries MJ, Anderson D, Williams L, Rieger R, Tunquist B, Walker D. ARRY-520 Combined With Pomalidomide Displays Enhanced Anti-Tumor Activity In Preclinical Models Of Multiple Myeloma. Blood. 2013;122(21):3167
- [Result] Petrelli NJ, Winer EP, Brahmer J, Dubey S, Smith S, Thomas C, Vahdat LT, Obel J, Vogelzang N, Markman M, Sweetenham JW, Pfister D, Kris MG, Schuchter LM, Sawaya R, Raghavan D, Ganz PA, Kramer B. Clinical Cancer Advances 2009: major research advances in cancer treatment, prevention, and screening--a report from the American Society of Clinical Oncology. J Clin Oncol. 2009 Dec 10;27(35):6052-69. doi: 10.1200/JCO.2009.26.6171. Epub 2009 Nov 9. No abstract available. PMID 19901123
- [Result] Kumar SK, Rajkumar SV, Dispenzieri A, Lacy MQ, Hayman SR, Buadi FK, Zeldenrust SR, Dingli D, Russell SJ, Lust JA, Greipp PR, Kyle RA, Gertz MA. Improved survival in multiple myeloma and the impact of novel therapies. Blood. 2008 Mar 1;111(5):2516-20. doi: 10.1182/blood-2007-10-116129. Epub 2007 Nov 1. PMID 17975015
- [Result] Richardson PG, Sonneveld P, Schuster MW, Irwin D, Stadtmauer EA, Facon T, Harousseau JL, Ben-Yehuda D, Lonial S, Goldschmidt H, Reece D, San-Miguel JF, Blade J, Boccadoro M, Cavenagh J, Dalton WS, Boral AL, Esseltine DL, Porter JB, Schenkein D, Anderson KC; Assessment of Proteasome Inhibition for Extending Remissions (APEX) Investigators. Bortezomib or high-dose dexamethasone for relapsed multiple myeloma. N Engl J Med. 2005 Jun 16;352(24):2487-98. doi: 10.1056/NEJMoa043445. PMID 15958804
- [Result] Singhal S, Mehta J, Desikan R, Ayers D, Roberson P, Eddlemon P, Munshi N, Anaissie E, Wilson C, Dhodapkar M, Zeddis J, Barlogie B. Antitumor activity of thalidomide in refractory multiple myeloma. N Engl J Med. 1999 Nov 18;341(21):1565-71. doi: 10.1056/NEJM199911183412102. PMID 10564685
- [Result] Dimopoulos M, Spencer A, Attal M, Prince HM, Harousseau JL, Dmoszynska A, San Miguel J, Hellmann A, Facon T, Foa R, Corso A, Masliak Z, Olesnyckyj M, Yu Z, Patin J, Zeldis JB, Knight RD; Multiple Myeloma (010) Study Investigators. Lenalidomide plus dexamethasone for relapsed or refractory multiple myeloma. N Engl J Med. 2007 Nov 22;357(21):2123-32. doi: 10.1056/NEJMoa070594. PMID 18032762
- [Result] Weber DM, Chen C, Niesvizky R, Wang M, Belch A, Stadtmauer EA, Siegel D, Borrello I, Rajkumar SV, Chanan-Khan AA, Lonial S, Yu Z, Patin J, Olesnyckyj M, Zeldis JB, Knight RD; Multiple Myeloma (009) Study Investigators. Lenalidomide plus dexamethasone for relapsed multiple myeloma in North America. N Engl J Med. 2007 Nov 22;357(21):2133-42. doi: 10.1056/NEJMoa070596. PMID 18032763
- [Result] Milross CG, Mason KA, Hunter NR, Chung WK, Peters LJ, Milas L. Relationship of mitotic arrest and apoptosis to antitumor effect of paclitaxel. J Natl Cancer Inst. 1996 Sep 18;88(18):1308-14. doi: 10.1093/jnci/88.18.1308. PMID 8797771
- [Result] Oltersdorf T, Elmore SW, Shoemaker AR, Armstrong RC, Augeri DJ, Belli BA, Bruncko M, Deckwerth TL, Dinges J, Hajduk PJ, Joseph MK, Kitada S, Korsmeyer SJ, Kunzer AR, Letai A, Li C, Mitten MJ, Nettesheim DG, Ng S, Nimmer PM, O'Connor JM, Oleksijew A, Petros AM, Reed JC, Shen W, Tahir SK, Thompson CB, Tomaselli KJ, Wang B, Wendt MD, Zhang H, Fesik SW, Rosenberg SH. An inhibitor of Bcl-2 family proteins induces regression of solid tumours. Nature. 2005 Jun 2;435(7042):677-81. doi: 10.1038/nature03579. Epub 2005 May 15. PMID 15902208
- [Derived] Ocio EM, Motllo C, Rodriguez-Otero P, Martinez-Lopez J, Cejalvo MJ, Martin-Sanchez J, Blade J, Garcia-Malo MD, Dourdil MV, Garcia-Mateo A, de Arriba F, Garcia-Sanz R, de la Rubia J, Oriol A, Lahuerta JJ, San-Miguel JF, Mateos MV. Filanesib in combination with pomalidomide and dexamethasone in refractory MM patients: safety and efficacy, and association with alpha 1-acid glycoprotein (AAG) levels. Phase Ib/II Pomdefil clinical trial conducted by the Spanish MM group. Br J Haematol. 2021 Feb;192(3):522-530. doi: 10.1111/bjh.16788. Epub 2020 Jun 5. PMID 32501528
- See also: Pethema Foundation — http://www.sehh.es/es/servicios-para-los-socios/pethema.html